CLINICAL TRIAL: NCT06214754
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial of the Efficacy and Safety of Intravascular High-pressure Cutting Balloon Catheters for PCI
Brief Title: Efficacy and Safety of Intravascular High-pressure Cutting Balloon Catheters for PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BM-839
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Atherosclerotic Plaque
MeSH Terms: conditions — Plaque, Atherosclerotic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravascular high-pressure cutting balloon catheter (Active Comparator)
  Interventions: Procedure: PCI
- Boston Scientific Corporation (Active Comparator)
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — The subjects underwent immediate coronary angiography after Percutaneous transluminal coronary angioplasty to evaluate the success rate of instruments, and immediate coronary angiography after PCI to evaluate the success rate of clinical treatment

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of intravascular high-pressure cut balloon catheter compared to cut balloon catheter during PCI, and to support product registration and clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 80 years of age (including boundary values) and have a life expectancy of more than 12 months；
2. Be able to understand the purpose of the study, voluntarily participate in and sign the informed consent, and be able and willing to accept the follow-up established in this study;
3. Ischemic cardiomyopathy with single or multiple coronary artery lesions and diagnostic evidence [e.g., stable angina, unstable angina, or occult ischemia (evidence of myocardial ischemia)；
4. Investigator is believed that the target atherosclerotic plaque needs to be incised and that predilation (if necessary) can enable the incised balloon to pass through the lesion；
5. The presence of coronary artery stenosis confirmed by imaging examination, suitable for percutaneous coronary intervention, coronary vessel stenosis ≥70%; Or ≥50% (visual) with evidence of ischemia, TIMI ≥ level 1；
6. The patient had autogenous coronary angiogenesis or restenosis, requiring stent treatment；
7. The reference vessel diameter of target lesion was 2.0mm-4.0mm, and the lesion length was ≤20mm；
8. When there are multiple lesions that need to be treated, only one in situ coronary lesion is selected as the target lesion, and the non-target lesion must be located on different vascular branches；

Exclusion Criteria:

1. Patients with bleeding tendencies, contraindications to antiplatelet and anticoagulant therapy, who are unable to undergo anticoagulant therapy；
2. Have had any myocardial infarction within a week；
3. People who have an allergic reaction to contrast media or can't take medication
4. There was severe renal failure with or without dialysis, glomerular filtration rate (eGFR) <30ml/min/1.73m2 or serum creatinine level >2.0 mg/ dl；
5. cardiogenic shock；
6. Patients who have received heart transplants；
7. Patients who are not eligible for coronary artery bypass surgery；
8. The patient had active peptic ulcer or active gastrointestinal bleeding within 1 month before surgery；
9. The patient had a stroke or transient ischemic attack within 2 months before surgery；
10. Patients in the pregnancy or lactation period；
11. Participants are currently participating in any other clinical trial within 1 month prior to the trial；
12. Patients deemed unsuitable for inclusion by other investigators；
13. Severe calcified lesions and twisted lesions or lesion sites > 45 degrees angled；
14. Lesions with significant endometrial tears
15. Unprotected left main lesion；
16. The contrast showed a blood clot；
17. Scaffold fracture lesion；
18. Distal stent lesion after stent implantation；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Device Procedural Success Rate | immediately after PTCA
  In the case of balloon dilatation and stenosis, balloon delivery, balloon filling and dilatation, balloon withdrawal pressure retraction and successful balloon retraction can be successfully completed. After balloon dilatation, residual stenosis of the target lesion is less than 50%

SECONDARY OUTCOMES:
Clinical Success Rate | immediately after PCI
  The residual lumen stenosis of the target lesion after surgery was less than 20%, the TIMI blood flow was grade 3, and there were no Major Adverse Cardiovascular Events during the follow-up period. MACE included cardiac death, myocardial infarction of the target vessel, or revascularization of the target lesion.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - the First Affiliated Hospital of USTC, Hefei, Anhui
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - the second affiliated hospital of Nanchang university, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Jilin, Jilin
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Neimenggu
  - First Affiliated Hospital of the Air Force Medical University, Xi'an, Shaanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan